CLINICAL TRIAL: NCT04655729
Title: Detection of Serum Protein Biomarkers to Predict and Monitor Response to Infliximab Using SOMAscan
Brief Title: Biomarkers to Predict and Monitor Response to Infliximab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Harland S. Winter, MD, Director, Pediatric IBD Program, Massachusetts General Hospital
Other Study IDs: 2019p002322
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SOMAscan analysis Inflammatory bowel disease serum biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Infliximab — Blood collection

SUMMARY:
The aim of the study is to generate novel minimally-invasive serum protein signatures and biomarkers in children and adolescents with Crohn's Disease (CD) that correlate with and can predict and monitor patients who will have a prolonged response to Infliximab so that personalized medicine can be applied to patients with CD.

DETAILED DESCRIPTION:
Prospective, observational study will enroll 120 unique pediatric Crohn's disease patients between the ages of 3-20 years among multiple sites. Patients will be naïve to TNF inhibitor. If patient is going to start infliximab or infliximab biosimilar, patient may be enrolled in study. Study length will be from commencement of infliximab until the infusion visit given at least 1 year after initiation. During the study, if the patient fails infliximab or biosimilar, they will be complete study once failure is indicated and discontinued on infliximab or biosimilar. Patients may be on concurrent IBD therapy such as antibiotics, mesalamines, immunomodulators and may continue in study if non-standard induction schedule or changes made during induction or maintenance to dose or frequency. Excluded patients will be those receiving infliximab or biosimilar infusions at home due to need for blood collection at time of infusion, on systemic corticosteroids (topical preparations such as budesonide are allowed), and those who have already undergone significant bowel surgery relating to their Crohn's.

Study visits will take place in conjunction with previously scheduled routine clinic visits or infusion visits. At initial study visit, demographics, medical and surgical history, PARIS classification, PCDAI, weight and height, fecal calprotectin, labs, EGD and colonoscopy report and pathology report, cross-sectional imaging reports and concurrent medications will be obtained and entered. Parameters measured at each study visit will include any obtained labs, weight and height, PARIS classification, PCDAI, infliximab dose (mg/kg) and dose interval. There will be four study visits throughout the course of 1 year after initiating infliximab. At these four visits, blood will be obtained in PAXgene tubes for RNA analysis and serum for banking for SOMAscan analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 3-20 years old
* Patient starting infliximab or infliximab biosimilar,
* Patients naïve to TNF inhibitor

Exclusion Criteria:

* Patients receiving infliximab or biosimilar infusions at home
* Patients already undergone significant bowel surgery relating to their Crohn's.

Ages: 3 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients 3-20 years old diagnosed with Crohn's Disease starting infliximab
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Define pretreatment serum protein biomarkers that predict and monitor response to TNF inhibitors (Discovery Cohort) | 2 years
  Run 120 pediatric Crohn's patients' serum at baseline, week 14, and week 54 on SOMAscan; Develop predictor model for protein biomarkers that predict response from baseline serum

SECONDARY OUTCOMES:
Identify pathophysiological mechanisms associated with response or lack of response in patients receiving IFX using SOMAscan. | 2 years
  Identify pathophysiological mechanisms associated with response or lack of response in patients receiving IFX using SOMAscan.
Use systems biology to map out pathways activated in those patients at week 14 that have clinical and laboratory response to infliximab | 2 years
  Use systems biology to map out pathways activated in those patients at week 14 that have clinical and laboratory response to infliximab

CONTACTS AND LOCATIONS:
Locations (1):
- MassGeneral for Children, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No